CLINICAL TRIAL: NCT05032768
Title: The Association Between Radiation Dermatitis and Skin Microbiome in Breast Cancer Patients Receiving Radiation After Mastectomy and Reconstructive Surgery
Brief Title: The Association Between Radiation Dermatitis and Skin Microbiome in Breast Cancer Patients
Status: Recruiting | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: FDRT-BC015
Record Dates: First submitted 2021-07-25; First posted 2021-09-02 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Radiation Dermatitis; Skin Microbiome; Breast Cancer; Reconstructive Surgery
MeSH Terms: conditions — Radiodermatitis; Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The skin microbiome will be collected and analyzed. Bacteria 16S rRNA amplicon sequencing and fungal rRNA its (internal transcribed spacer) sequencing will be used to analyze skin microorganisms (including bacteria and fungi)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Severe radiation dermatitis: RTOG/EORTC grade 2 and above
  Interventions: Radiation: post-operative radiotherapy
- No or mild radiation dermatitis: RTOG/EORTC grade 0 or 1
  Interventions: Radiation: post-operative radiotherapy

INTERVENTIONS:
Radiation: post-operative radiotherapy — Breast cancer patients who have received reconstructive surgery will receive post-operative radiotherapy.

SUMMARY:
The breast cancer patients who received radiotherapy after mastectomy and breast reconstruction will be enrolled. The skin microbiome before radiotherapy and its changes after radiotherapy will be analyzed systematically to find out whether the skin microbiome is associated with the severity of radiation dermatitis.

DETAILED DESCRIPTION:
Radiotherapy is an important treatment for breast cancer patients. About 95% of patients receiving radiotherapy will develop a degree of radiation dermatitis. Radiation dermatitis is usually limited to the site of radiation treatment. Symptoms vary and can range from itching, burning and pain to open or bleeding ulcers, which can greatly affect the quality of life of patients. Severe acute radiation dermatitis can lead to interruption or delay of treatment. At present, there is no standard for the prevention and treatment of radiation dermatitis. Our skin is home to millions of bacteria, fungi and viruses which compose the skin microbiota. Skin microbiota interacts with skin and affects physiology and immunity of the skin. Previous studies have reported the effects of radiotherapy on skin and immune system. However, so far, no studies have analyzed the effects of radiotherapy on skin microbiome and how skin microbiome affects the skin immune responses after radiotherapy. In this study, the breast cancer patients who received radiotherapy after mastectomy and breast reconstruction will be enrolled. The skin microbiome before radiotherapy and its changes after radiotherapy will be analyzed systematically to find out whether the skin microbiome is associated with the severity of radiation dermatitis. The long-term goal of this study is to deepen the understanding of the role of skin microbiome in the occurrence and development of radiation dermatitis, and provide a basis for subsequent exploration to reduce radiation dermatitis by regulating skin microecology.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients
2. Invasive breast cancer confirmed by pathology
3. Underwent mastectomy and breast reconstruction
4. Radiotherapy after breast reconstruction
5. ECOG score 0-1
6. Signed informed consent

Exclusion Criteria:

1. Previous breast or chest radiotherapy
2. Other serious skin diseases (systemic lupus erythematosus, skin sclerosis, et al) and cannot receive radiotherapy
3. Pregnant women
4. Patients who are unwilling or unable to receive regular follow-up.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who have underwent mastectomy and breast reconstruction and who will receive post-operative radiotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Skin microbiome differences between patients with and without >=2 acute radiation dermatitis | 3 months
  Acute radiation dermatitis will be graded per the Toxicity Criteria of the Radiation Therapy Oncology Group (RTOG)

SECONDARY OUTCOMES:
Skin microbiome differences between patients with and without >=2 late radiation dermatitis | 5 years
  Late radiation dermatitis will be graded per the Toxicity Criteria of the Radiation Therapy Oncology Group (RTOG)

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, MD, Ph.D, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided